CLINICAL TRIAL: NCT01014728
Title: Comparison of Intraoperative Bleeding During Endoscopic Sinus Surgery Between Patients Receiving Total Intravenous Anesthesia With Propofol and Patients Receiving an Inhalational Anesthetic With Sevoflurane
Brief Title: Intraoperative Bleeding During Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-317A
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Results first posted 2014-01-09 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous anesthesia (Active Comparator): Intravenous anesthesia with propofol for endoscopic sinus surgery
  Interventions: Drug: propofol
- Inhalation anesthesia (Active Comparator): Inhalation anesthesia with sevoflurane for endoscopic sinus surgery
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: propofol — 100-200mcg/kg/min by infusion
  Arms: Intravenous anesthesia
Drug: sevoflurane — 1-3% of sevoflurane (expired)
  Arms: Inhalation anesthesia

SUMMARY:
The purpose of this study is to compare the blood loss during sinus surgery looking at two different types of anesthesia: either intravenous anesthesia with propofol or inhalational anesthesia with sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients who are 18 years of age or older,
* ASA grade 1 (normal otherwise healthy patient),
* ASA grade 2 (patient with mild systemic disease),
* patients who have chronic sinusitis with or without nasal polyps.

Exclusion Criteria:

* pregnancy,
* abnormal coagulation panel
* preoperative use of NSAIDS or ASA medications within 7 days,
* end-stage renal disease,
* allergy to any of the used medications,
* maximal body mass index over 35

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Anesthesia: After induction, the intravenous anesthesia group received an infusion of propofol (100-200 μg/kg/min) for endoscopic sinus surgery.
- Inhalation Anesthesia: After induction, the inhalation anesthesia group received sevoflurane (1% to 3%) for endoscopic sinus surgery.
Period: Overall Study
Arm/Group | Intravenous Anesthesia | Inhalation Anesthesia
Started | 18 | 15
Completed | 18 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Anesthesia | Inhalation Anesthesia | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (16.9) | 43.4 (16.6) | 42.3 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Estimated Blood Loss
Description: Estimated blood loss in milliliters per hour is calculated by subtracting the volume of total irrigation used during the case from the total amount of fluid in the suction canister at the end of surgery and dividing by surgical time in hours.
Time Frame: from the start of surgery to the end of surgery, up to 6 hours
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Intravenous Anesthesia | Inhalation Anesthesia
Number analyzed (Participants) | 18 | 15
mL/h | 78.5 (59.4) | 80.3 (70.2)
Statistical Analysis 1: Comparison: Intravenous Anesthesia vs Inhalation Anesthesia; Test type: Superiority or Other; p = 0.937, t-test, 2 sided

2. Secondary Outcome: Anesthesiologist Numeric Rating Scale (ANRS)
Description: The anesthesiologist numeric rating scale is to rate the ease of the anesthesia technique ranging from 0 to 10 (10 is best, 0 is worst).
Time Frame: at the end of surgery (up to 6 hours)
Population: There were three patients in the inhalation anesthesia group with missing values.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Intravenous Anesthesia | Inhalation Anesthesia
Number analyzed (Participants) | 18 | 12
units on a scale | 7.25 [2 to 10] | 9 [8 to 10]
Statistical Analysis 1: Comparison: Intravenous Anesthesia vs Inhalation Anesthesia; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Surgeon's Numeric Rating Scale (SNRS)
Description: The surgeon's numeric rating scale(SNRS)is to rate the surgical conditions (mucosal bleeding and visibility) on a scale ranging from 0 to 10, with 0 defined as cadaveric conditions and 10 as severe bleeding requiring constant suction.
Time Frame: at the end of surgery (up to 6 hours)
Population: There were three patients in the inhalation anesthesia group with missing values.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Intravenous Anesthesia | Inhalation Anesthesia
Number analyzed (Participants) | 18 | 12
units on a scale | 6 [5 to 9] | 7.25 [4 to 10]
Statistical Analysis 1: Comparison: Intravenous Anesthesia vs Inhalation Anesthesia; Test type: Superiority or Other; p = 0.461, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Intravenous Anesthesia | Inhalation Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15
Other Adverse Events (participants affected / at risk) | 0/18 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No